CLINICAL TRIAL: NCT02437019
Title: An Early Access Program (EAP) for Ibrutinib (PCI-32765) in Subjects With Relapsed or Refractory Chronic Lymphocytic Leukemia (CLL)
Brief Title: Early Access Program (EAP) for Ibrutinib in Participants With Relapsed or Refractory Chronic Lymphocytic Leukemia (CLL)
Status: Approved for marketing | Type: Expanded Access
Sponsor: Janssen-Cilag Farmaceutica Ltda. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR106344; 54179060CLL3005 (Other: Janssen-Cilag Farmaceutica Ltda.)
Record Dates: First submitted 2015-04-17; First posted 2015-05-07 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: B-cell Chronic Lymphocytic Leukemia
Keywords: PCI-32765; Ibrutinib; Early access program; Chronic lymphocytic leukemia; Relapsed or refractory chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence | interventions — ibrutinib

INTERVENTIONS:
Drug: PCI-32765 (Ibrutinib) — Participants will receive PCI-32765 (ibrutinib) 420 mg (three 140-mg capsules) oral once daily continuously on a 28-day cycle.

SUMMARY:
The purpose of this study is to provide early access to Ibrutinib treatment for participants with relapsed or refractory Chronic Lymphocytic Leukemia (CLL) and collect additional safety data while the medication is not commercially available.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), multi-center (when more than one hospital or medical school team work on a medical research study) early access program (EAP) study. The study will be conducted in 2 phases: a Screening Phase (approximately 30 days prior to administration of first dose) and a Program Drug Phase (Day 1 up to 30 Days after last dose of study drug). Enrolled participants will receive 420 milligram (mg) oral ibrutinib once daily on a 28-day cycle until disease progression, occurrence of unacceptable toxicity, no longer achieving clinical benefit, or the end of program. Treatment will be continuous (without interruption) and self-administered. Disease evaluations will be conducted according to local standard of care as clinically indicated. Participant's safety will be monitored throughout the study. All enrolled and on-going participants in the program will continue to receive ibrutinib by the EAP until marketing approval or 6 months after this date.

ELIGIBILITY:
Inclusion Criteria:

* Has Eastern Cooperative Oncology Group (ECOG) performance status of less than (<) 2
* Has a diagnosis of Chronic Lymphocytic Leukemia (CLL) that meets published diagnostic criteria (Hallek 2008):

  1. Monoclonal B-cells (either kappa or lambda light chain restricted) that are clonally co-expressing at least one B-cell marker (Cluster of Differentiation 19 [CD19], CD20, or CD23) and CD5
  2. The diagnosis of CLL requires a history of lymphocytosis with a B-lymphocyte count greater than or equal to (>=) 5,000/microliter (μl)
* Active disease meeting at least one of the International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2008 criteria
* Must have received at least one prior therapy for CLL and not be appropriate for treatment or retreatment with purine analog based therapy
* Able to receive all outpatient treatment and all laboratorial monitoring at the institution that administers program drug

Exclusion Criteria:

* Known central nervous system (CNS) lymphoma or leukemia
* Known prolymphocytic leukemia or history of or currently suspected Richter's transformation
* Uncontrolled autoimmune hemolytic anemia (AIHA) or idiopathic thrombocytopenic purpura (ITP)
* Prior exposure to ibrutinib or randomization in an ibrutinib study
* Requires treatment with a strong Cytochrome P3A4/5 (that is, CYP3A4/5) Inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Farmaceutica Ltda. Clinical Trial, Study Director — Janssen-Cilag Farmaceutica Ltda.
Locations (6):
- Brazil (6):
  - Barretos
  - Florianópolis
  - Fortaleza
  - Porto Alegre
  - Rio de Janeiro
  - São Paulo